CLINICAL TRIAL: NCT06384664
Title: Cryoablation Effects on Acute and Chronic Pain After Thoracotomy and Thoracoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Rishindra Reddy, Research Professor of Thoracic Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00241242
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Intrathoracic Procedure
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryosurgery; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intercostal nerve block (Active Comparator): Standard of care
  Interventions: Procedure: Standard of Care
- Cryoablation (Experimental): Cryoablation is a procedure that is used to freeze and burn away tissue cells via a device called a cryosphere which emits a freezing gas.
  Interventions: Device: Atricure's crysoSPHERE probe

INTERVENTIONS:
Device: Atricure's crysoSPHERE probe — Cryoablation is a procedure that is used to freeze and burn away tissue cells via a device called a cryosphere which emits a freezing gas.
  Other Names: cryoablation
  Arms: Cryoablation
Procedure: Standard of Care — An intercostal nerve block involves injecting anesthetic medications into nerves around the thoracic incision to provide temporary longer term pain relief after surgery.
  Other Names: Intercostal nerve block
  Arms: Intercostal nerve block

SUMMARY:
The researchers will compare the common methods of post-surgical pain control, such as epidural or intercostal nerve block with a newer method called cryoablation. The research team is conducting this study to determine if cryoablation provides more effective pain control when compared to an epidural or intercostal nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients who could receive cryoablation in an elective open thoracic (posterolateral thoracotomy) or minimally invasive (thoracoscopy, including robotic) procedures at Michigan Medicine
* Patient is opioid naïve

Exclusion Criteria:

* Patients who are pregnant
* Patients with cognitive impairment
* Patients with psychological disorders
* Patients with prior thoracic surgery
* Patients with fibromyalgia
* Patients with redo ipsilateral thoracic surgery
* Patients undergoing bilateral thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Severity of pain in the peri-operative period | Post-op day 1 and day of hospital discharge, approximately 3 days
  Pain measured using a numeric rating scale ranging from 1-10 where a higher pain score indicates more pain severity
Inflammatory cytokine levels as measured by blood samples | Pre-surgery, 6-hours after end of surgery and 24-hours after surgery
  Levels are measured using blood sample collection and assay specifically assessing IL-1, IL-6, TNF-a
Inflammatory cytokines (IL-1, IL-6, TNF-a) levels correlations to pain score | Pre-surgery, 6-hours after end of surgery and 24-hours after surgery
  Correlations with the pain scores from outcome #1
Peri-operative pain scores between different surgical incisions (posterolateral thoracotomy vs thoracoscopy) | baseline (pre-op), post-op day 1, day of hospital discharge, approximately 3 days, 2-weeks postop and 30-, 90-, and 180-days postop
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) pain intensity surveys
Peri-operative nerve function between different surgical incisions (posterolateral thoracotomy vs thoracoscopy) | baseline (pre-op), post-op day 1, day of hospital discharge, approximately 3 days, 2-weeks postop and 30-, 90-, and 180-days postop
  assessment of feeling or touching sensations along the thoracic cavity measured using dermatone assessment

SECONDARY OUTCOMES:
Quality of life score as measured by SF-36 Health questionnaire | baseline (prior to surgery), day of hospital discharge, approximately 3 days, 30-days, 90-days and 180-days post-op.
  36 item survey instrument
Cost (including postoperative epidural management, narcotic pain medication, and outpatient pain management) | Up to 180-days postop
  Hospital charges for cases that get standard of care postop pain management versus cases that receive cryoablation.
Workflow/time | Up to 180-days postop
  Including items such as length of operating room use and length of hospital stay

OTHER OUTCOMES:
Complications following surgery | Up to 180-days following surgery
  Any unexpected or unanticipated incidents, symptoms or medical issues following surgery
Length of stay | Up to hospital discharge, approximately 3 days
  length of hospital stay
Time to ambulation | Up to 180-days following surgery
  Day of first ambulation documented
Chronic Pain medication use through 6 months | Up to 180-days after surgery
Chronic pain through 6 months. | Up to 180-days after surgery
  Chronic pain is defined as pain that lasts for over three months as assessed by the PROMIS Pain Intensity survey
Chronic pain through 6 months. | Up to 180-days after surgery
  Chronic pain is defined as pain that lasts for over three months as assessed by the PROMIS Pain Interference survey
Chronic pain through 6 months. | Up to 180-days after surgery
  Chronic pain is defined as pain that lasts for over three months as assessed by the PROMIS Neuropathic Pain Quality Survey
Incentive spirometry volumes in the peri-operative period (POD 1 and 2) | Postop day 1 and 2
Oxygen requirement | Up to 180-days postop
  documentation of oxygen use
Hospital charges and hospital reimbursement by different payors | Up to 180-days postop

CONTACTS AND LOCATIONS:
Overall Officials: Rishindra Reddy, MD, MBA, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No